CLINICAL TRIAL: NCT01008969
Title: Practice Procedure for 99mTc-Sulfur Nanocolloid Lymphatic Drainage Mapping in Prostate Cancer Using SPECT-CT (Single Photon Emission Computed Tomography / Computed Tomography)
Brief Title: Feasibility of Using SPECT/CT Imaging to Map Lymphatic Drainage Patterns in Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC085513, H46038-33934
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer
Keywords: Prostate; SPECT/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: SPECT-CT imaging — SPECT/CT for 3-dimensional mapping of 99mTc-sulfur nanocolloid in order to identify personalized lymphatic drainage patterns

SUMMARY:
The purpose of this study is to develop a practice procedure for lymphatic drainage mapping with the intent of providing a new tool that could potentially be used for radiation treatment planning. High-risk prostate cancer patients who are scheduled to be treated with intensity-modulated radiotherapy (IMRT) may be eligible to enroll in this study. 99mTc-sulfur nanocolloid, a radiopharmaceutical ("tracer") will be injected by a urologist using transrectal ultrasound guidance (TRUS)at the UCSF Urology Clinic. Participants will then undergo SPECT/CT imaging at the UCSF Nuclear Medicine Clinic. This study will evaluate the feasibility of transporting patients to the Nuclear Medicine Clinic for imaging within 1-3 hours after administration of 99mTc-sulfur nanocolloid.

DETAILED DESCRIPTION:
The entire study procedure involves 1) preparation of 99mTc-sulfur nanocolloid, 2) administration of 99mTc-sulfur nanocolloid with transrectal ultrasound guidance, 3) transfer of the patient to the Nuclear Medicine clinic for SPECT/CT (Infinia Hawkeye, GE Healthcare) imaging, and 4) tomographically capturing distributions of 99mTc-sulfur nanocolloid uptake in the patient's lymphatic drainage sites within a practical image acquisition time (1-3 h postinjection) considering the patient transit time between injection and imaging.

Administration of 99mTc-sulfur nanocolloid will be performed at the UCSF Urology clinic. The injection will be performed following the clinically accepted method that has been described by European investigators. 99mTc-sulfur nanocolloid imaging utilizes trace amounts of radioactivity. 100-200 MBq (2.7-5.4 mCi) of 99mTc-sulfur nanocolloid will be administered into two lobes of the prostate gland under transrectal ultrasound guidance with three fractions each into peripheral and central zone of the prostatic apex, mid portion, and base. 1% Lidocaine may be administered for local anesthesia per routine clinical protocol as deemed appropriate by the performing urologist.

The procedure will be considered feasible if the practice procedure (from injection to completion of imaging) is successfully implemented within 3 hours of injection (including patient transport time). Imaging will be considered successful if radiotracer is qualitatively detected within the prostate and local lymphatic system.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥ 18 years
* Diagnosis of definitive high-risk prostate cancer
* Clinically eligible and scheduled for definitive IMRT treatment with pelvic lymph nodal radiation (not a study procedure)
* At least one of the following risk factors:

  1. Pathologically confirmed pelvic nodal involvement;
  2. Enlarged pelvic lymph nodes (greater than 1 cm in the short axis) visible on CT or MRI images, or
  3. Greater than 15% risk of lymph node involvement calculated using the equation: Risk of positive nodes (%) = (2/3) prostate specific antigen (PSA) + [(Gleason score - 6)] × 10]. This formula is used to estimate the pathologic stage of prostate cancer with preoperative prostate specific antigen (PSA) and Gleason score, and adopted by many radiation oncology clinics, including our own radiation oncology physicians.
* Ability to give written informed consent and willingness to comply with the requirements of the protocol

Exclusion Criteria:

• Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youngho Seo, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 99mTc-sulfur Nanocolloid SPECT/CT: SPECT/CT imaging of administered 99mTc-sulfur nanocolloid within 3 hours after injection in patients with prostate cancer
Period: Overall Study
Arm/Group | 99mTc-sulfur Nanocolloid SPECT/CT
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 99mTc-sulfur Nanocolloid SPECT/CT
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Successfully Completed 99mTc-sulfur Nanocolloid SPECT/CT Within 3 Hours After Injection
Description: Successful completion of 99mTc-sulfur nanocolloid SPECT/CT means that the images were obtained within 3 hours, and the images showed patients' lymphatic drainage.
Time Frame: 1 day
Population: We reviewed the imaging results of this procedure by SPECT/CT. Percentage of participants who received SPECT/CT scans of 99mTc-sulfur nanocolloid was analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- 99mTc-sulfur Nanocolloid SPECT/CT: There was only one arm for this study. All participants who had prostate cancer received 99mTc-sulfur nanocolloid injection and imaged by SPECT/CT within 3 hours of injection.
Arm/Group | 99mTc-sulfur Nanocolloid SPECT/CT
Number analyzed (Participants) | 10
Percentage of Participants | 100

2. Secondary Outcome: Percentage of Images With Detectable Sentinel Lymph Nodes (LNs) From 99mTc-sulfur Nanocolloid SPECT/CT Scans
Description: There was only one arm for this study. All participants who had prostate cancer received 99mTc-sulfur nanocolloid injection and imaged by SPECT/CT within 3 hours of injection. The imaging studies qualitatively detected radiotracer distribution within the prostate and local lymphatic system. The detection of the radiotracer distribution was performed by experienced attending nuclear medicine physicians at UCSF. The qualitative detection includes visual lymph node uptake seen by SPECT scans overlaid on coregistered CT scans.
Time Frame: 1 day
Population: We reviewed the imaging results of this procedure by SPECT/CT. We calculated the percentage of images with detectable lymph nodes from SPECT/CT images in these participants.
Measure: Number; unit: percentage of images identifying LNs
Arm/Group | 99mTc-sulfur Nanocolloid SPECT/CT
Number analyzed (Participants) | 10
percentage of images identifying LNs | 100

ADVERSE EVENTS:
Time Frame: One week. One-week adverse event assessment was about the SPECT/CT imaging procedure as well as the radiotracer injection.
Description: The adverse event assessment was performed by verbal communication with the participants.
Arm/Group | 99mTc-sulfur Nanocolloid SPECT/CT
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No